CLINICAL TRIAL: NCT04358614
Title: Baricitinib Therapy in COVID-19: A Pilot Study on Safety and Clinical Impact
Brief Title: Baricitinib Therapy in COVID-19
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fabrizio Cantini (Other)
Responsible Party: Sponsor-Investigator, Fabrizio Cantini, MD, Head of Rheumatology Department, Principal investigator, Hospital of Prato
Organization: Hospital of Prato (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HPrato-4
Record Dates: First submitted 2020-04-19; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: COVID; Pneumonia
Keywords: COVID-19; BARICITINIB; MODERATE DISEASE
MeSH Terms: conditions — Pneumonia; COVID-19 | interventions — baricitinib; Lopinavir; Ritonavir; BID protein, human

STUDY DESIGN:
Intervention Model Description: Baricitinib treated patients compared with controls (previously COVID-19 receving standard therapy)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case patients (Active Comparator): Consecutive patients with COVID moderate pneumonia treated with baricitinib tablets 4 mg/day
  Interventions: Drug: Baricitinib 4 MG Oral Tablet
- Controls (Other): Consecutive patients with COVID moderate pneumonia treated with standard therapy before the date of the first baricitinib-treated patient.
  Interventions: Drug: Baricitinib 4 MG Oral Tablet

INTERVENTIONS:
Drug: Baricitinib 4 MG Oral Tablet — Baricitinib+antiviral therapy administration for 2 weeks
  Other Names: Lopinavir/Ritonavir tablets 250 mg/bid

SUMMARY:
Retrospective study on the efficacy of baricitinib in 12 COVID-19 patients with moderate pneumonia.

DETAILED DESCRIPTION:
Baricitinib, an anti-Janus kinase inhibitor (anti-JAK) acting against JAK1 and JAK2 that inhibits JAK1- and JAK2-mediated cytokine release, was recently described using BenevolentAI's proprietary artificial intelligence-derived knowledge graph, as an agent that reduces the endocytosis into target cells, and to inhibit the entry. Based on its potential action on inhibition of SARS-CoV-2 entry, and on its known effects on reduction of cytokine release, baricitinib therapy was proposed in patients with moderate pneumonia to explore: the safety of this drug combined with antiviral (lopinavir-ritonavir) in COVID-19; as second outcome, to evaluate the impact of baricitinib in terms of clinical, laboratory, respiratory parameters, and reduction of ICU admission.

Baricitinib was combined with antivirals because it does not interact with them due to its prevalent renal elimination.

ELIGIBILITY:
Inclusion Criteria:

* SARS-Co-V2 positivitity to the nasal-swab by reverse-transcriptase-polymerase chain- reaction (RT-PCR) assay tested by the local diagnostic laboratory
* Age >18 and <85 years
* Presence of at least 3 of the following symptoms as present fever, cough, myalgia, fatigue.
* Presence of radiological findings of pneumonia assessed by chest radiograph, computed tomography, or pulmonary ultrasound.
* Peripheral capillary oxygen saturation (SpO2) > 92% on room air at screening
* PaO2/FiO2 >100-300 mmHg at arterial blood gas analysis.

Exclusion Criteria:

* Age < 18 and >85
* History of thrombophlebitis
* Latent tuberculosis infection (based on the positivity to QuantiFERON Plus positivity, Qiagen, Germany)
* Pregnancy and lactation
* History of malignancies over the previous 5 years, current diagnosis of malignancy
* Inability or unwillingness to sign a written consent.
* Transaminases values 4-fold higher than the upper normal limit.
* HBV and HCV positivity.
* Current Herpes zoster infection.
* Evidence of concomitant bacterial infections.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety of baricitinib combined with antiviral (lopinavir-ritonavir) in terms of serious or non-serious adverse events incidence rate. | 2 weeks
  All adverse event recording

SECONDARY OUTCOMES:
To evaluate the impact of baricitinib in terms of clinical, laboratory, respiratory parameters. | 2 weeks
  The percentage of patients improving the clinical and respiratory parameters compared with controls.
ICU admission rate | 2 weeks
  The percentage of ICU admission in baricitinib group as compared with controls.
Discharge rate. | 2 weeks
  The percentage of discharged in baricitinib group as compared with controls.

CONTACTS AND LOCATIONS:
Locations (1):
- Fabrizio Cantini, Prato, Tuscany, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Conner SD, Schmid SL. Identification of an adaptor-associated kinase, AAK1, as a regulator of clathrin-mediated endocytosis. J Cell Biol. 2002 Mar 4;156(5):921-9. doi: 10.1083/jcb.200108123. Epub 2002 Mar 4. PMID 11877461
- [Background] Ferner RE, Aronson JK. Chloroquine and hydroxychloroquine in covid-19. BMJ. 2020 Apr 8;369:m1432. doi: 10.1136/bmj.m1432. No abstract available. PMID 32269046
- [Background] Richardson P, Griffin I, Tucker C, Smith D, Oechsle O, Phelan A, Rawling M, Savory E, Stebbing J. Baricitinib as potential treatment for 2019-nCoV acute respiratory disease. Lancet. 2020 Feb 15;395(10223):e30-e31. doi: 10.1016/S0140-6736(20)30304-4. Epub 2020 Feb 4. No abstract available. PMID 32032529
- [Background] Stebbing J, Phelan A, Griffin I, Tucker C, Oechsle O, Smith D, Richardson P. COVID-19: combining antiviral and anti-inflammatory treatments. Lancet Infect Dis. 2020 Apr;20(4):400-402. doi: 10.1016/S1473-3099(20)30132-8. Epub 2020 Feb 27. No abstract available. PMID 32113509
- [Background] Subbe CP, Kruger M, Rutherford P, Gemmel L. Validation of a modified Early Warning Score in medical admissions. QJM. 2001 Oct;94(10):521-6. doi: 10.1093/qjmed/94.10.521. PMID 11588210